CLINICAL TRIAL: NCT06659666
Title: Opportunities to Optimize COPD Management Using the COPD Optimiser Online Tool in Dutch General Practice
Brief Title: The COPD Optimiser
Status: Completed | Type: Observational
Sponsor: General Practitioners Research Institute (Network)
Collaborators: AstraZeneca (Industry)
Responsible Party: Sponsor
Other Study IDs: GPRI_2024_003
Record Dates: First submitted 2024-10-22; First posted 2024-10-26 (Actual); Last update posted 2025-12-26 (Actual); Status verified 2025-12

CONDITIONS: COPD
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Usual care COPD consultation with the COPD Optimiser: Primary care patients with a current COPD diagnosis who visit the GP team for their COPD are eligible to participate in the study. Patients with COPD will be recruited from 10-15 primary care practices in the Netherlands. The population includes men and women ≥35 years of age with clinically diagnosed COPD. The diagnosis of COPD is allowed to be a clinical diagnosis rendered by a member of the GP team, without the requirement to conduct additional confirm- atory testing. Furthermore, a limited number of in- and exclusion criteria will be adopted, to make sure the research population closely resembles the real world.
  Interventions: Device: COPD Optimiser

INTERVENTIONS:
Device: COPD Optimiser — Patients will receive enhanced usual medical care as determined by their physician. The study visit is a standard consultation supported by the COPD Optimiser webtool. The extra elements added to the COPD consultation are the use of the COPD Optimiser and a short questionnaire directly following the consultation on the patient's experience with the COPD Optimiser. Patients can additionally consent to two optional elements: 1) a determination of blood eosinophil count using a point of care test and 2) a brief interview on their experience with the COPD Optimiser. this tool creates an overview of fac- tors and characteristics that may be associated with suboptimal COPD and provides GOLD guideline-based management suggestions. Implementation of the COPD Optimiser will sup- port healthcare professionals in providing optimal care for their COPD patients by providing individualized GOLD-guided management suggestions.

SUMMARY:
Rationale: The Global Initiative for Chronic Obstructive Lung Disease (GOLD) report pro- vides clinical treatment guidelines for COPD aimed at relieving and reducing the impact of symptoms, and reducing the risk of adverse health events, such as exacerbations. Despite the availability of these COPD treatment guidelines, evidence suggests that available thera- pies may not be utilized to their full potential to optimize disease management and outcomes for patients. So far, there is a lack of knowledge on the optimalisation opportunities of patients with COPD in a primary care setting.

Objective: The primary objective is to describe the GOLD-guided management suggestions obtained from the COPD Optimiser, in order to gain insight into optimalisation opportunities in a Dutch primary care population of patients with COPD.

Study design: This is a non-interventional prospective observational study, taking place in a real-world primary care setting.

Study population: Patients diagnosed with COPD are eligible to participate. A limited number of in- and exclusion criteria will be adopted, to make sure the research population closely resembles the real world.

ature and extent of the burden and risks associated with participation, benefit and group relatedness: Study specific involvement is limited to the one visit for the participant. Participants will receive enhanced usual medical care as determined by their physician and will not be randomly allocated to an experimental intervention or care as usual. The partici- pating general practices and participants in the study will be reimbursed for the time spent on this study. Risks of participating in the study are deemed to be negligible. All participants will use their own medication and follow the management plan that is in line with guidelines. The study specific additions to the consultation are administering a (not emotionally demanding) questionnaire and drawing a small amount of blood from the finger, to measure the level of blood eosinophils, using a point-of-care method. This is a test that may cause a slight incon- venience for the patient, although this test is less invasive than typical blood draws that would be part of the newest international guideline.

Primary objective

1. Describe the GOLD-guided management suggestions obtained from the COPD Optimiser, in order to gain insight into optimalisation opportunities in a Dutch primary care pop- ulation of patients with COPD. The endpoint for the primary objective is the number of times that each manage- ment suggestion was given

ELIGIBILITY:
Inclusion Criteria:

* Physician diagnosis of COPD (ICPC R95),
* Capacity to understand and provide written informed consent.

Exclusion Criteria:

* Active diagnosis of Asthma (ICPC R96)
* Patients participating in an interventional clinical trial

Min Age: 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Primary care patients with a current COPD diagnosis who visit the GP team for their COPD are eligible to participate in the study. Patients with COPD will be recruited from 10-15 primary care practices in the Netherlands. The population includes men and women ≥35 years of age with clinically diagnosed COPD. The diagnosis of COPD is allowed to be a clinical diagnosis rendered by a member of the GP team, without the requirement to conduct additional confirmatory testing. Furthermore, a limited number of in- and exclusion criteria will be adopted, to make sure the research population closely resembles the real world.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2024-10-09 (Actual); Primary Completion 2025-01-20 (Actual); Study Completion 2025-07-24 (Actual)

PRIMARY OUTCOMES:
patterns of co-occurrence of GOLD-guided management suggestions in a Dutch primary care population of patients with COPD. | Immediately after the procedure
  The primary endpoint is the number of times that each management suggestion was given. With this endpoint, we can describe the proportion of primary care patients with COPD of whom disease management can be optimized per GOLD-guided management suggestions from the COPD Optimiser. Incidence will be described for each of the possible management suggestions from the COPD Optimiser.

SECONDARY OUTCOMES:
Co-occurance and concordance of GOLD-based management suggestions | Immediately after the procedure
  The secondary study endpoints are
  1. The presence of co-occurring GOLD-guided management suggestions from the COPD Optimiser in primary care patients with COPD
  2. The proportion of patients for whom the current medication regimen is not in line with the GOLD pharmacological treatment recommendation, either:
     1. The proportion of patients that received a GOLD-guided step-up advice from the COPD Optimiser
     2. The proportion of patients that received a GOLD-guided step-down advice from the COPD optimiser

OTHER OUTCOMES:
User experience of healthcare providers & participants | Immediately after the procedure for SUS. For the exploratory interviews, through study completion, within 12 weeks of study end
  The endpoint for the user experience of the healthcare provider is captured by employing the System Usability Scale, adapted to Dutch (SUS-D). This questionnaire explores the perceived usefulness and ease of use of the tool. We will add questions about the likelihood to act upon the management suggestions from the COPD optimiser, as well as the likelihood to continue the use of the COPD optimiser in the future.
  For participants, the exploratory parameters are their experience during the visit (in comparison with previous COPD consultations) (e.g. duration, relevance of questions, actions after the consultation).

CONTACTS AND LOCATIONS:
Locations (2):
- Netherlands (2):
  - General practices in Netherlands, Groningen, Provincie Groningen
  - GPRI, Groningen, Provincie Groningen

IPD SHARING:
Plan to Share IPD: Undecided
This is currently under review

REFERENCES:
- See also: 2024 GOLD Report - Global Initiative for Chronic Obstructive Lung Disease - GOLD. Ac- cessed July 19, 2024. https://goldcopd.org/2024-gold-report/ — https://goldcopd.org/2024-gold-report/